CLINICAL TRIAL: NCT07085936
Title: Determinants of Stress and Stigma Among Caregivers of Psychiatric Patients: The Effect of a Video-Based Orientation Intervention and Feature Importance Analysis Using SVR
Brief Title: Stress and Stigma Among Psychiatric Caregivers: Effects of a Video-Based Orientation and Feature Importance Via SVR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Merve Aydın, Associate Profesor, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Stigma_Psychiatric Caregivers
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Family Members of Psychiatric Patients
Keywords: stigma; stress; anxiety
MeSH Terms: conditions — Social Stigma; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): First-degree relatives of psychiatric inpatients who receive a structure Video-based orientation program with four sessions over one week. Sessions cover stigma, mental illness education, and coping strategies, led by psychiatric nurses. Pre- and post-tests assess outcomes.
  Interventions: Behavioral: Video-based orientation program
- Control group (No Intervention): Participants receive standard verbal orientation routinely provided in the hospital, without structured sessions or video materials.

INTERVENTIONS:
Behavioral: Video-based orientation program — The intervention group will receive a structured video-based orientation program developed for first-degree relatives of psychiatric inpatients. The program consists of four sessions (each 45-60 minutes) delivered over one week by psychiatric nurses. Topics include an introduction to the psychiatric unit, understanding stigma, basic information on mental illnesses, and strategies for coping with stigma. Educational videos support learning and discussion. Unlike the control group, this intervention emphasizes stigma awareness and emotional support. Pre- and post-tests are used to assess perceived stress and stigma.
  Arms: Experimental Group

SUMMARY:
Determinants of Stress and Stigma Among Caregivers of Psychiatric Patients: The Effect of a Video-Based Orientation Intervention

Conducted by:

Faculty of Medicine, Karadeniz Technical University (KTU)

Purpose of the Study:

This study aims to examine the stress and stigma experienced by first-degree relatives (parent, spouse, or child) of patients hospitalized in a psychiatric unit, and to evaluate the effect of a video-based orientation training on these experiences.

Where and When Is the Study Conducted? The study will take place in the psychiatric ward of KTU Farabi Hospital between July 15 and September 30, 2025.

Who Can Participate?

You can take part in this study if you are:

A first-degree relative of a psychiatric inpatient,

18 years of age or older,

Able to read, write, and communicate verbally,

Willing to participate voluntarily.

What Will Happen During the Study?

Participants will be randomly assigned to one of two groups:

Intervention group: Will receive video-based orientation training.

Control group: Will receive standard routine orientation.

The video training includes four sessions (each lasting about 45-60 minutes). These sessions cover:

Introduction to the psychiatric unit and the research,

What stigma means and how it affects caregivers,

Basic information about mental illnesses and treatment,

How to understand and cope with stigma.

You will be asked to complete two short questionnaires: one before and one week after the training. These help us understand your stress levels and feelings of stigma.

Confidentiality and Ethics:

This study has been approved by the Scientific Research Ethics Committee of Karadeniz Technical University. All information you provide will be kept confidential and used only for scientific purposes. Your participation is voluntary, and you may withdraw from the study at any time without giving a reason.

Contact Information:

If you would like more information, feel free to contact the research team.

DETAILED DESCRIPTION:
Determinants of Stress and Stigma Among Caregivers of Psychiatric Patients: The Effect of a Video-Based Orientation Intervention and Feature Importance Analysis Using Support Vector Regression

Conducted by:Faculty of Medicine, Karadeniz Technical University (KTU)

Overview and Purpose of the Study:This scientific study is designed to explore the emotional and social challenges faced by family members who care for individuals with mental illness. In particular, it focuses on two common experiences: stress and stigma.

The goal is to assess whether a specially prepared video-based orientation training can help reduce the perceived stress levels and the feelings of being stigmatized among caregivers. By participating in this study, you will contribute to valuable research that can improve future support programs for families like yours.

What Is Stigma and Why Is It Important?"Stigma" refers to the negative beliefs and attitudes that society may hold about mental illness. Unfortunately, these beliefs do not only affect individuals with mental illness-they can also impact their families and caregivers. You may have experienced situations where people judged you or treated you differently because you care for someone with a psychiatric condition. This study aims to help reduce such experiences by offering accurate information, emotional support, and tools for coping.

Study Duration and Location:The study will be conducted between July 15 and September 30, 2025, at the psychiatric ward of KTU Farabi Hospital, located in northeastern Türkiye. This ward is a secure unit where patients with severe psychiatric symptoms receive treatment and support.

Who Can Participate?You are eligible to participate if you:

Are a first-degree relative (mother, father, spouse, or child) of a patient currently hospitalized in the psychiatric unit,

Are 18 years or older,

Can read, write, and communicate verbally,

Volunteer to participate in the study.

Individuals who have a current psychiatric diagnosis themselves or a history of substance use, dementia, or other serious mental conditions will not be included in the study.

What Does Participation Involve?

After agreeing to join the study, you will be randomly placed into one of two groups:

The Intervention Group: You will attend four video-supported orientation sessions.

The Control Group: You will receive routine orientation as typically provided in the hospital.

The video-based training program will be led by mental health professionals and held in a quiet, comfortable room within the psychiatric unit. Each session will last about 45-60 minutes, and will cover the following topics:

Introduction to the psychiatric unit and the research - a video tour and Q&A session

Understanding stigma - what stigma is, how it affects caregivers, and personal experiences

Basic information about mental illnesses - causes, symptoms, treatment options, and how to provide care

Coping with stigma - strategies and tools to manage emotional and social stress

You will also be asked to fill out two brief questionnaires:

Once before the training (pre-test)

Once one week after the training (post-test) These questionnaires help us evaluate the impact of the training on your stress and stigma levels.

Benefits of Participation:

Gain knowledge and insight about the mental health system and caregiving.

Learn new strategies to cope with emotional challenges and societal stigma.

Contribute to scientific research that may improve mental health care policies and family support services.

Confidentiality and Ethics:This study has been reviewed and approved by the Scientific Research Ethics Committee of Karadeniz Technical University. All the information you provide will be kept strictly confidential and used solely for research purposes. Participation is entirely voluntary, and you are free to withdraw at any time without any consequences.

Contact Information:If you have any questions or would like further details about the study, please feel free to contact the research team. Your questions are always welcome.

We thank you sincerely for considering participation in this important research.

ELIGIBILITY:
Inclusion Criteria: First-degree relatives (mother, father, spouse, or child) of patients admitted to the psychiatric inpatient unit

Age 18 years or older

Willing to participate voluntarily

Able to read and write, and to communicate verbally well enough to complete the study instruments -

Exclusion Criteria: Individuals with a current psychiatric diagnosis based on DSM-5 criteria

History of alcohol or substance use

Diagnosed with dementia or other organic mental disorders

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Parents' Internalized Stigma of Mental Illness Scale (PISMI) | Baseline (pre-test) and 1 week after intervention (post-test)
Parents' Internalized Stigma of Mental Illness Scale (PISMI) | Baseline (pre-test) and 1 week after intervention (post-test)
  The PISMI is a 29-item self-report instrument developed by Boyd-Ritsher et al. (2003) to measure internalized stigma in parents of individuals with mental illness. It includes five subscales: Alienation, Stereotype Endorsement, Perceived Discrimination, Social Withdrawal, and Resistance to Stigma. Items are rated on a 4-point Likert scale. Higher scores indicate greater levels of internalized stigma. The Turkish version was adapted by Gül Dikeç et al. (2019).

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS-14) | Baseline (pre-test) and 1 week after intervention (post-test)
  The PSS-14 is a 14-item self-report scale developed by Cohen et al. (1983) to measure the degree to which situations in one's life are appraised as stressful. Scores range from 0 to 56; higher scores indicate higher perceived stress. Turkish version validated by Eskin et al. (2013).

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical Univercity, Trabzon, Turkey (Türkiye)

DOCUMENTS (1):
  • Study Protocol (2025-07-18): https://cdn.clinicaltrials.gov/large-docs/36/NCT07085936/Prot_000.pdf